CLINICAL TRIAL: NCT05378503
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Phase IV Clinical Trial to Evaluate Efficacy and Safety of Qsymia in Obese Patients
Brief Title: Phase IV Study of Qsymia in Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-119
Record Dates: First submitted 2022-05-10; First posted 2022-05-18 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Obesity
Keywords: Obesity; Qsymia; Phentermine; Topiramate; Alvogen Korea
MeSH Terms: conditions — Obesity | interventions — Qsymia; Maintenance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active (Experimental): 1. Administration of Qsymia 3.75mg/23mg once a daily for 2-week(W2), and then administration of Qsymia 7.5mg/46mg once a daily for 12-week(W14).
  2-1. At W14, if the weight loss rate is 3% or more, administration of Qsymia 7.5mg/46mg once a daily by the end of visit(W56).
  2-2. At W14, if the weight loss rate is NOT 3% or more, administration of Qsymia 11.25mg/69mg once a daily for 2-week(W16), and then administration of Qsymia 15mg/92mg once a daily by the end of visit(W56).
  Interventions: Drug: Qsymia 3.75Mg-23Mg Extended Release Capsule; Drug: Qsymia 7.5Mg-46Mg Extended Release Capsule; Drug: Qsymia 11.25Mg-69Mg Extended Release Capsule; Drug: Qsymia 15Mg-92Mg Extended Release Capsule
- Placebo (Placebo Comparator): Administration of Qsymia placebo once a daily by the end of visit(W56).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Qsymia 3.75Mg-23Mg Extended Release Capsule — From W0 to W2, once a daily.
  Other Names: Low dose titration
  Arms: Active
Drug: Qsymia 7.5Mg-46Mg Extended Release Capsule — 1. From W2 to W14, once a daily.
  2. At W14, if the weight loss rate is 3% or more, from W14 to W56(the end of visit), once a daily.
  Other Names: Low dose maintenance
  Arms: Active
Drug: Qsymia 11.25Mg-69Mg Extended Release Capsule — At W14, if the weight loss rate is NOT 3% or more, from W14 to W16, once a daily.
  Other Names: High dose titration
  Arms: Active
Drug: Qsymia 15Mg-92Mg Extended Release Capsule — At W14, if the weight loss rate is NOT 3% or more, from W16 to W56(the end of visit), once a daily.
  Other Names: High dose maintenance
  Arms: Active
Drug: Placebo — From W0(Randomisation) to W56(the End of visit) once a daily.
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to evaluate the weight loss effect and safety after administration of the test drug Qsymia in obese patients.

To this end, the primary objective is to compare the weight change rate (%) between the study groups compared to the placebo groups at week 56 after administration of the investigational product.

The secondary objective is to compare the weight change rate (%) at each evaluation point after administration of the investigational product, the proportions of subjects who lost more than 5% and more than 10% of weight at each evaluation point, and changes in weight/BMI/waist circumference/heart rate/blood pressure between the study groups compared to the placebo groups.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women aged 19 to 70 years
2. Obese patients with BMI ≥ 25 kg/m2 at screening visit and visit 2
3. Those who agreed to low-calorie regimen and exercise therapy during the study at screening visit
4. From screening visit prior to randomization visit (Visit 2), low-calorie regimen and exercise therapy compliances are all ≥ 70%
5. From screening visit prior to randomization visit (Visit 2), those who fails to lose weight by at least 10% due to a low-calorie regimen and exercise therapy.
6. Those who voluntarily decided to participate and gave written consent after being provided with and understanding the detailed explanation on this clinical trial

Exclusion Criteria:

1. Patients with glaucoma
2. Thyroid dysfunction (hyperthyroidism, hypothyroidism) (however, for hypothyroidism, the case of taking therapeutic agents stably at least 3 months prior to the screening visit is allowed)
3. Arteriosclerosis patients with symptoms such as intermittent lameness and lower extremity pain
4. Patients with type 1 diabetes or those with type 2 diabetes who are taking diabetic medications other than metformin. (However, metformin is allowed only if it was administered without dose change 1 month prior to screening visit.)
5. Those who are taking monoamine oxidase (MAO) inhibitors at screening visit or who had taken less than 14 days before screening
6. Patients with SBP ≥ 160 mmHg, DBP ≥ 100 mmHg, or pulmonary hypertension at screening visit
7. A history of eating disorders, drug or alcohol abuse
8. A history of surgery for weight loss (e.g., bariatric surgery)
9. A weight change of > 5kg within 3 months prior to the screening visit
10. A history of mental illness (e.g., bipolar disorder, depression, suicidal ideation, etc.)
11. Obesity due to endocrine disorders or genetic obesity
12. A history of kidney stones or gallbladder stones within 6 months of the screening visit
13. Patients who need to take furosemide (loop diuretic) or hydrochlorothiazide (thiazide-like diuretic) during the study (However, it is allowed only if it is administered for treatment of hypertension without dose change 3 months prior to screening visit.)
14. Patients with renal impairment (CrCl < 60 mL/min)
15. Patients with hepatic impairment (AST, ALT ≥ 2.5 X ULN)
16. A history of treatment for transient ischemic attack (TIA), myocardial infarction, unstable angina, cerebral infarction, and cerebral hemorrhage, or angioplasty or coronary artery bypass grafting within 6 months prior to the screening visit (if it occurs before 6 months and is currently stable, it is possible to enroll)
17. Patients with severe heart failure (NYHA class III or higher), arrhythmia requiring treatment, and clinically significant heart valve disease
18. A history of anaphylaxis to active or minor ingredients of the investigational product
19. Hypersensitivity reaction or idiosyncrasy to sympathomimetic amine
20. A history of malignant tumor within 5 years prior to the screening visit (Surgery-resected basal cell carcinoma of the skin or squamous cell carcinoma of the skin or cervical intraepithelial neoplasia or thyroid cancer with no evidence of recurrence after 3 years of surgery are allowed)
21. Pregnant or lactating women
22. Those who disagree to the use of a medically acceptable contraception (see Section 14.1) during the study
23. A history of systemic steroid administration for 14 days or more within 3 months of screening visit
24. Within 3 months prior to the screening visit

    * Taking Qsymia or
    * Taking phentermine and topiramate in combination for weight loss or
    * Taking phentermine or topiramate for other purposes
25. Taking other appetite suppressants (including herbal medicines) excluding Qsymia (or drugs containing active ingredient of Qsymia) within 6 months prior to the screening visit
26. Participation in other clinical trials within 3 months before the screening visit (participation is based on the last administration date of the investigational product)
27. Other cases where the investigator determined that the subject is ineligible for participation in the obesity clinical study based on the history of medical or surgical disease or laboratory test results

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Weight change rate(percent) | Week 56
  Weight change rate(percent) from the baseline at week 56 after administration of the investigational product.

SECONDARY OUTCOMES:
Weight change rate(percent) | weeks 14, 28, and 42
  Weight change rate(percent) from the baseline at weeks 14, 28, and 42 after administration of the investigational product.
The proportions(percent) of subjects whose body weight has changed | weeks 14, 28, 42, and 56
  The proportions(percent) of subjects whose body weight has changed by 5 percents or more and 10 percents or more at weeks 14, 28, 42, and 56 after administration of the investigational product.
The amounts of changes from the baseline in body weight | weeks 14, 28, 42, and 56
  The amounts of changes from the baseline in body weight at weeks 14, 28, 42, and 56 after administration of the investigational product
The amounts of changes from the baseline in waist circumference | weeks 14, 28, 42, and 56
  The amounts of changes from the baseline in waist circumference at weeks 14, 28, 42, and 56 after administration of the investigational product
The amounts of changes from the baseline in BMI | weeks 14, 28, 42, and 56
  The amounts of changes from the baseline in BMI at weeks 14, 28, 42, and 56 after administration of the investigational product
The amounts of changes from the baseline in heart rate | weeks 14, 28, 42, and 56
  The amounts of changes from the baseline in heart rate at weeks 14, 28, 42, and 56 after administration of the investigational product
The amounts of changes from the baseline in blood pressure(Systolic and diastolic) | weeks 14, 28, 42, and 56
  The amounts of changes from the baseline in blood pressure(Systolic and diastolic) at weeks 14, 28, 42, and 56 after administration of the investigational product

OTHER OUTCOMES:
The amounts of changes from the baseline in body composition (visceral fat area) | weeks 14, 28, 42, and 56
  (Optional) The amounts of changes from the baseline in body composition (visceral fat area) at weeks 14, 28, 42, and 56 after administration of the investigational product
The amounts of changes from the baseline in body composition (body fat percentage) | weeks 14, 28, 42, and 56
  (Optional) The amounts of changes from the baseline in body composition (body fat percentage) at weeks 14, 28, 42, and 56 after administration of the investigational product
The amounts of changes from the baseline in blood lipids (TC, TG, HDL-C, LDL-C) | weeks 14, 28, 42, and 56
  The amounts of changes from the baseline in blood lipids (TC, TG, HDL-C, LDL-C) at weeks 14, 28, 42, and 56 after administration of the investigational product
The amounts of changes from the baseline in diabetes indicators (HbA1c) | weeks 14, 28, 42, and 56
  The amounts of changes from the baseline in diabetes indicators (HbA1c) at weeks 14, 28, 42, and 56 after administration of the investigational product
The amounts of changes from the baseline in diabetes indicators (FBS) | weeks 14, 28, 42, and 56
  The amounts of changes from the baseline in diabetes indicators (FBS) at weeks 14, 28, 42, and 56 after administration of the investigational product
The amounts of changes from the baseline in diabetes indicators (Fasting Insulin) | weeks 14, 28, 42, and 56
  The amounts of changes from the baseline in diabetes indicators (Fasting Insulin) at weeks 14, 28, 42, and 56 after administration of the investigational product
The amounts of changes from the baseline in diabetes indicators (HOMA-IR) | weeks 14, 28, 42, and 56
  The amounts of changes from the baseline in diabetes indicators (HOMA-IR) at weeks 14, 28, 42, and 56 after administration of the investigational product

CONTACTS AND LOCATIONS:
Overall Officials: ChangBeom Lee, M.D., Ph.D., Principal Investigator — Hanyang Univ. Guri Hospital
Locations (8):
- South Korea (8):
  - KyungHee Univ. Hospital, Seoul, Dongdaemun-gu
  - KyungHee Univ. Hospital at Gangdong, Seoul, Gangdong-gu
  - The Catholic Univ. of Korea Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Sejong Hospital, Bucheon-si, Gyeonggi-do
  - Hanyang Univ. Guri Hospital, Guri-si, Gyeonggi-do
  - Gil Hospital, Incheon, Namdong-gu
  - GangNeung Asan Hospital, Gangneung, Sacheon-myeon
  - Severance Hospital, Seoul, Seodaemun-gu

IPD SHARING:
Plan to Share IPD: No
Confidential